CLINICAL TRIAL: NCT07359612
Title: Improving Sleep Health Through Magnesium Supplementation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 54246
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sleep Health
Keywords: nutrition, sleep, magnesium
MeSH Terms: interventions — Magnesium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnesium 250 mg (Experimental): Participants will consume 250mg of magnesium supplement daily over a 56-day period.
  Interventions: Dietary Supplement: Magnesium 250 mg

INTERVENTIONS:
Dietary Supplement: Magnesium 250 mg — Participants will consume 250 mg of magnesium once a day preferably with a meal

SUMMARY:
Research has shown that there is a close relationship between sleep and diet. It has been shown that a vitamin and mineral rich diet is related to better sleep. This relationship can go both ways as poor sleep can also impact on your diet. Specifically, low magnesium levels have been associated with insomnia and adding magnesium to the diet of an individual with insomnia can help with their symptoms. Whilst this is known about insomnia, far less is known about the impact of magnesium on general sleep health. In other words, people who don't have a sleep disorder but could be sleeping better generally.

The aim of this study is to determine whether supplementing with Magnesium in those people who are deficient over a period of 8 weeks improves overall sleep health.

DETAILED DESCRIPTION:
This study will be an open label trial 60 participants will consume 250mg of magnesium supplement daily over a 56-day period. During their participation in this study participants will visit the Sleep Lab on three (3) occasions to pick up or drop off an actiwatch and receive the supplement (visit 2).

Informed consent will be obtained online and be followed by an online demographic screener, sleep screener (SDSCL-25), chronotype screener (MCTQ, HO), standard health screener and 3-day food diary.

On visit 1 participants will receive an actiwatch and undergo a 7 night sleep monitoring period where remote assessment of sleep via Actigraphy watch will be completed (baseline).

On visit 2, 7-10 days following visit 1, participants will arrive at the lab return their actigraphy watch and be provided with a new actiwatch and the supplement. Participants will provide a detailed recall of their diet in the past 24 hours and complete a Gastrointestinal symptoms questionnaire - The questionnaire asks 11 questions, plus a 12th open-ended question, about gastrointestinal experiences, with 5 possible ratings: 'not at all' (score of 0), 'A little' (score of 1), 'a moderate amount' (score of 2), 'quite a lot' (score of 3) and 'a severe amount' (score of 4). Scores can range between 0-44 with a higher score indicating a more negative experience of symptoms.

On visit 3, 56 days following, visit 2, participants will return the actiwatch and any supplements left over then be debriefed and participant payment details will be taken to facilitate their participant payment (£50).

Note: Timings given here are approximates for illustrative purposes and may be subject to change due to unexpected delays.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adult between the ages of 18 and 39 years of age.
* Have a stable sleep/wake schedule (bedtime between 9pm and 1am and wake time between 6am and 10am at least 5 nights per week)
* Are a fluent English speaker
* Diet which is low in magnesium
* Self-identify as a poor sleeper (i.e. poor sleep quality or unrefreshing sleep).

Exclusion Criteria:

* Have symptoms of COVID-19
* Display evidence of current or recent sleep disorders (e.g. sleep apnea, insomnia, circadian rhythm disorders); an initial screening for sleep disorders will be conducted using the Sleep Disorders Screening Checklist - 25 (SDS-CL). Have a history of seizures or epilepsy
* Have recently (within the last 12 weeks) had an infection and/or used antibiotic medication
* Are pregnant, seeking to become pregnant or lactating
* Are a shift worker or a recent history of shift work in the previous 6 months
* Are participating in other intervention research trials
* Have experienced travel across multiple time zones within the last three months or will be experiencing travel across multiple time zones during the study.
* Have recently been diagnosed and/or treated for a mental health or substance use disorder.
* Are currently unwell with anything that impacts sleep.
* Are taking any medication which has a sedative effect
* Are currently using medication which affects the central nervous system.
* Are currently misusing alcohol or drugs.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Actigraphy - Sleep onset latency | Change from baseline following 56 days of supplement consumption
  recorded minutes taken from intention to sleep to sleep initiation
Sleep Diary -Sleep Latency | Change from baseline following 56 days of supplement consumption
  how long, in minutes, the individual felt it took them to fall asleep after intending to sleep
Actigraphy - total sleep time | Change from baseline following 56 days of supplement consumption
  recorded minutes asleep over entire sleep period
Sleep Diary - total sleep time | Change from baseline following 56 days of supplement consumption
  how long, in minutes, the individual reports being asleep during the night between initiation and termination of sleep, accounting for nocturnal wake periods
Actigraphy - Wake after sleep onset (WASO) | Change from baseline following 56 days of supplement consumption
  recorded minutes awake during the entire sleep period following sleep onset
Sleep Diary - Wake After Sleep Onset (WASO) | Change from baseline following 56 days of supplement consumption
  how long, in minutes, the individual reports being awake during the night after sleep initiation
Actigraphy - Sleep efficiency | Change from baseline following 56 days of supplement consumption
  ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed (percentage)
Sleep Diary - Sleep efficiency | Change from baseline following 56 days of supplement consumption
  Total Sleep Time divided by Time in Bed x 100, expressed as a percentage
Dietary assessment- 7 day dietary recall | Change from baseline following 56 days of supplement consumption
  Participants will complete 7 day dietary recall questionnaire
Gastrointestinal symptoms questionnaire | Change from baseline following 56 days of supplement consumption
  When completing the assessment, participants will answer in relation to their experiences in the previous 7 days. The questionnaire asks 11 questions, plus a 12th open-ended question, about gastrointestinal experiences, with 5 possible ratings; 'not at all' (score of 0), 'A little' (score of 1), 'a moderate amount' (score of 2), 'quite a lot' (score of 3) and 'a severe amount' (score of 4). Scores can range between 0-44 with a higher score indicating a more negative experience of symptoms
Generalized Anxiety Disorder 7- Item Scale scores (GAD-7) | Change from baseline following 56 days of supplement consumption
  The GAD-7 is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. It contains 7 items with answers ranging from "Not at all" to "Nearly every day".
Patient Health Questionnaire (PHQ9) | Change from baseline following 56 days of supplement consumption
  The PHQ9 will screen for depression symptoms. It is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression: It incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool.

SECONDARY OUTCOMES:
Munich Chronotype Questionnaire (MCTQ) | Change from baseline following 56 days of supplement consumption
  Self-rated scale to assess individual phase of entrainment on work and work-free days, developed in ages 6 to > 65 years; tool to collect primary sleep times, such as bed- and rise-times, plus the clock time of becoming fully awake as well as sleep latency and inertia, in addition to other time points and rate themselves as one of the seven chronotypes.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria Sleep Research, Northumbria University, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: No